CLINICAL TRIAL: NCT05009147
Title: Effects of Manual Massage on Improving Behavioral and Psychological Symptoms of Dementia and Sense of Burden Among Caregivers
Brief Title: Home-based Massage by Caregivers for Dementia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taipei University of Nursing and Health Sciences (Other)
Responsible Party: Principal Investigator, CY Song, Prof, National Taipei University of Nursing and Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: CTH-109-2-5-025
Record Dates: First submitted 2021-08-08; First posted 2021-08-17 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2022-04

CONDITIONS: Dementia; Massage; Burden
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): receive whole body manual massage
  Interventions: Other: Home-based massage by caregivers for dementia
- control group (No Intervention): After experiment, receive whole body manual massage

INTERVENTIONS:
Other: Home-based massage by caregivers for dementia — A total of 40 patients with dementia and their family caregivers will be included and randomly allocated to experiment (n=20) or control group (n=20). The experiment and control group will receive whole body manual massage and placebo intervention (30 minutes once per week for 8 continuous weeks), respectively.
  Arms: experimental group

SUMMARY:
The purpose of this study is to investigate the effects of manual massage on improving behavioral and psychological symptoms of dementia and sense of burden among caregivers.

DETAILED DESCRIPTION:
A total of 40 patients with dementia and their family caregivers will be included and randomly allocated to experiment (n=20) or control group (n=20). The experiment and control group will receive whole body manual massage and placebo intervention (30 minutes once per week for 8 continuous weeks), respectively.

ELIGIBILITY:
Inclusion Criteria:

* Over 65 years old, diagnosed with dementia, agitation or depression, irregular massage and exercise habits.

Exclusion Criteria:

* Those who have open wounds, inflammation, infection, burns and scalds, artificial blood vessels in the hands, or diagnosed as inappropriate for massage in the near future, the severity of symptoms affects the study participants.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-05-31 (Estimated); Study Completion 2022-05-31 (Estimated)

PRIMARY OUTCOMES:
change agitation | before , during and after 8-weeks massage training interventions
  Cohen-Mansfield Agitation Inventory (CMAI)
change depression | before , during and after 8-weeks massage training interventions
  Cornell Scale for Depression in Dementia (CSDD)
change stress | before , during and after 8-weeks massage training interventions
  Perceived Stress Scale(PSS)

CONTACTS AND LOCATIONS:
Overall Officials: Chen-Yi Song, Principal Investigator — National Taipei University of Nursing and Health Sciences
Locations (1):
- National Taipei University of Nursing and Health Sciences, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided